CLINICAL TRIAL: NCT01678131
Title: A Randomized Clinical Trial Using Fine Needle Aspiration For Evaluation of Hepatic Pharmacokinetics of MK-7009 in Chronic Hepatitis C Patients
Brief Title: Evaluating Fine Needle Aspiration to Measure Hepatic Vaniprevir (MK-7009) Concentrations in Participants With Chronic Hepatitis C (MK-7009-048)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7009-048; 2012-003284-21 (EudraCT Number)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — vaniprevir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaniprevir 600 mg (Experimental): Participants received 600 mg vaniprevir only on days 1-7, and had postdose liver biopsy done by FNA and CNB from Day 7 up to Day 10.
  Interventions: Drug: Vaniprevir 600 mg; Procedure: Liver samples from FNA; Procedure: Liver samples from CNB
- Vaniprevir 600 mg + Peg-IFN + RBV (Experimental): Participants received 600 mg vaniprevir on Days 1-7; Peg-IFN alpha-2b once a week, RBV daily from Day 1 up to Day 21; and had postdose liver biopsy done by FNA and CNB from Day 7 up to Day 10.
  Interventions: Drug: Vaniprevir 600 mg; Biological: Peg-IFN alfa-2b; Biological: Ribavirin; Procedure: Liver samples from FNA; Procedure: Liver samples from CNB
- Vaniprevir 300 mg + Peg-IFN + RBV (Experimental): Participants received 300 mg vaniprevir from Days 1-7; Peg-IFN alpha-2b once a week, RBV daily from Day 1 up to Day 21; and had postdose liver biopsy done by FNA and CNB from Day 7 up to Day 10.
  Interventions: Biological: Peg-IFN alfa-2b; Biological: Ribavirin; Procedure: Liver samples from FNA; Drug: Vaniprevir 300 mg; Procedure: Liver samples from CNB

INTERVENTIONS:
Drug: Vaniprevir 600 mg — Vaniprevir capsules, were administered orally, twice per day (BID) to achieve a final daily dose of 600 mg on Days 1 through 6; and a single dose of 600 mg, orally, on Day 7.
  Other Names: MK-7009
  Arms: Vaniprevir 600 mg; Vaniprevir 600 mg + Peg-IFN + RBV
Biological: Peg-IFN alfa-2b — Peg-IFN alfa-2b was administered at 1.5 µg/kg per week by subcutaneous injections on Days 1, 8, 15 and 21
  Other Names: PegIntron™
  Arms: Vaniprevir 300 mg + Peg-IFN + RBV; Vaniprevir 600 mg + Peg-IFN + RBV
Biological: Ribavirin — Ribavirin capsules were administered on Days 1-21, orally, twice daily for a total daily dose of 600 - 1400 mg, depending on the participant's weight
  Other Names: Rebetol™
  Arms: Vaniprevir 300 mg + Peg-IFN + RBV; Vaniprevir 600 mg + Peg-IFN + RBV
Procedure: Liver samples from FNA — Liver samples were collected from Day 7 up to Day 10 by FNA at 3 of 5 specified postdose timepoints.
Drug: Vaniprevir 300 mg — Vaniprevir capsules were administered orally, twice per day to achieve a final daily dose of 300 mg on Days 1 through 6; and a single dose of 300 mg, orally, on Day 7.
  Other Names: MK-7009
  Arms: Vaniprevir 300 mg + Peg-IFN + RBV
Procedure: Liver samples from CNB — Liver samples were collected from Day 8 up to Day 10 by CNB at 1 of 3 specified postdose timepoints.

SUMMARY:
This study will evaluate the technical feasibility of using fine needle aspiration (FNA) of liver tissue to obtain vaniprevir (MK-7009) liver pharmacokinetic (PK) data, working towards identifying a minimally invasive, reproducible platform to measure liver PK. The study will be done in 2 parts. In Part 1, participants will be randomized to one of five FNA/core needle biopsy (CNB) time-point collection sequences. In Part 2, participants will be randomized to one of two possible doses of vaniprevir and will be assigned to one of five FNA/CNB time-point collection sequences; participants in Part 2 will also receive background therapy with pegylated interferon alpha-2b (Peg-IFN alpha-2b) and ribavirin (RBV). The primary hypothesis is that there is a greater than 80% posterior probability that vaniprevir concentrations are successfully obtained at least 60% of the time from FNA liver samples collected at 2 of 3 specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥18.5 kg/m^2 and ≤32.0 kg/m^2
* Under evaluation for treatment of chronic hepatitis C virus (HCV)
* Chronic compensated, genotype 1 HCV infection
* Treatment-naïve or previously treated and tolerated at least 12 weeks of continuous licensed interferon (including pegylated interferon) and ribavirin combination therapy with at least a partial response, or previously treated with investigational products and/or vaccines, other than HCV nonstructural proteins (NS) NS3/4A protease inhibitors, either alone or in combination with other licensed therapies
* Able to avoid use of anticoagulants, nonsteroidal anti-inflammatory agents and aspirin for at least seven (7) days preceding the initial liver biopsy and continuing throughout the entire study
* Female participants of childbearing potential or male participants with female sexual partners of childbearing potential must agree to use two acceptable methods of birth control from 2 weeks prior to the first dose through at least 6 months after last dose of study drug, or longer if dictated by local regulation

Exclusion criteria:

* Pregnant, lactating, or intending to become pregnant or donate eggs, or intending to donate sperm
* History of stroke, chronic seizures, or major neurological disorder
* Did not achieve a viral response to prior treatment with licensed interferon-based therapy
* Previously treated with an NS3/4A protease inhibitor (investigational or licensed)
* Evidence or history of chronic hepatitis not caused by HCV infection including but not limited to non-HCV viral hepatitis, nonalcoholic steatohepatitis (NASH), drug-induced hepatitis or autoimmune hepatitis
* Clinical or laboratory evidence of cirrhosis or other advanced liver disease
* Decompensated liver disease as indicated by a history of ascites, hepatic encephalopathy, or bleeding esophageal varices
* Diagnosed with or suspected of having hepatocellular carcinoma
* Co-infection with human immunodeficiency virus (HIV)
* Positive hepatitis B surface antigen or other evidence of active hepatitis B infection
* History of gastric bypass surgery or bowel resection
* History of clinically significant uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of clinically significant neoplastic disease
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL], wine [125 mL], or distilled spirits [25 mL]) per day
* Regular user, including use of any illicit drugs, or has a history of drug (including alcohol) abuse within the last 3 months
* Surgery or donation of 1 unit of blood (approximately 500 mL) or participation in another investigational study within a period of 4 weeks prior to the prestudy (screening) visit
* History of multiple and/or severe allergies, or has had an anaphylactic reaction or intolerability to prescription or nonprescription drugs or food

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2013-08-27 (Actual); Study Completion 2013-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gao W, Webber AL, Maxwell J, Anderson M, Caro L, Chung C, Miltenburg AMM, Popa S, Van Dyck K, Wenning L, Mangin E, Fandozzi C, Railkar R, Shire NJ, Fraser I, Howell B, Talal AH, Stoch SA. Fine-Needle Aspiration for the Evaluation of Hepatic Pharmacokinetics of Vaniprevir: A Randomized Trial in Patients With Hepatitis C Virus Infection. Clin Pharmacol Ther. 2020 Jun;107(6):1325-1333. doi: 10.1002/cpt.1737. Epub 2020 Feb 8. PMID 31868916
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-048&kw=7009-048&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 mg Vaniprevir: Participants received 600 mg vaniprevir only from Days 1-7; and had postdose liver biopsy from Day 7 up to Day 10 done by Fine Needle Aspiration (FNA) and Core Needle Biopsy (CNB).
- 300 mg Vaniprevir + PegIFN/RBV: Participants received 300 mg vaniprevir from Days 1-7; Pegylated Interferon (Peg-IFN) alpha-2b once weekly, Ribavirin (RBV) twice daily from Day 1 up to Day 21; and had postdose liver biopsy from Day 7 up to Day 10 done by FNA and CNB.
- 600 mg Vaniprevir + PegIFN/RBV: Participants received 600 mg vaniprevir from Days 1-7; Peg-IFN once weekly, RBV twice daily from Day 1 up to Day 21; and had postdose liver biopsy from Day 7 up to Day 10 done by FNA and CNB.
Period: Overall Study
Arm/Group | 600 mg Vaniprevir | 300 mg Vaniprevir + PegIFN/RBV | 600 mg Vaniprevir + PegIFN/RBV
Started | 10 | 10 | 11
Completed | 10 | 9 | 9
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg Vaniprevir | 300 mg Vaniprevir + PegIFN/RBV | 600 mg Vaniprevir + PegIFN/RBV | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (10.6) | 43.9 (12.1) | 38.9 (8.0) | 42.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 9 | 8 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Whom Detectable Concentrations of Hepatic Vaniprevir Are Obtained by FNA
Description: Liver samples were collected by FNA at 3 of 5 of the following specified postdose timepoints: 3, 12, 24, 48 and 72 hours after a single vaniprevir dose on Day 7. The technical success of the FNA procedure was established for a participant if vaniprevir was detected from at least 2 of the 3 FNA collection timepoints.
Time Frame: Day 7 up to Day 10 at 3 of the following timepoints: 3, 12, 24, 48 and 72 hours postdose
Population: Participants treated with vaniprevir who had hepatic FNA collected at 3 timepoints. One participant from the 300 mg Vaniprevir + Peg-IFN/RBV treatment group, and one participant from the 600 mg Vaniprevir + Peg-IFN/RBV treatment group discontinued treatment prior to collection of 3 FNAs, and were therefore excluded from the analysis.
Measure: Number; unit: Participants
Groups:
- 600 mg Vaniprevir: Participants received 600 mg vaniprevir only from Days 1-7; and had postdose liver biopsy from Day 7 up to Day 10 done by FNA and CNB.
Arm/Group | 600 mg Vaniprevir | 300 mg Vaniprevir + PegIFN/RBV | 600 mg Vaniprevir + PegIFN/RBV
Number analyzed (Participants) | 10 | 9 | 10
Participants | 10 | 9 | 10
Statistical Analysis 1: Comparison: 600 mg Vaniprevir vs 300 mg Vaniprevir + PegIFN/RBV vs 600 mg Vaniprevir + PegIFN/RBV; The posterior percentage probability of the true success rate of the FNA procedure for the 3 combined treatment groups (n=29) was determined by a Bayesian calculation, using a Jeffrey's prior distribution (i.e. Beta [0.5,0.5]) on the true success rate. Neither P-values, nor confidence intervals are estimated in this analysis. The primary hypothesis was met if the posterior percentage probability was > 80% that the true success rate is at least 60%; Test type: Superiority or Other; Posterior Percentage Probability = 100

ADVERSE EVENTS:
Time Frame: up to 14 days after last treatment with vaniprevir (up to approximately Day 21)
Arm/Group | 600 mg Vaniprevir | 300 mg Vaniprevir + PegIFN/RBV | 600 mg Vaniprevir + PegIFN/RBV
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 10/10 | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg Vaniprevir (N=10) | 300 mg Vaniprevir + PegIFN/RBV (N=10) | 600 mg Vaniprevir + PegIFN/RBV (N=11)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 4 (4)
Fever (General disorders) | 0 (0) | 10 (17) | 8 (10)
Rigors (General disorders) | 0 (0) | 1 (1) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 5 (6)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.